CLINICAL TRIAL: NCT04826224
Title: A Pilot Study For The Use Of Human Autologous Bone Marrow Aspirate Concentrate (BMAC) Combined With Arthroscopic Surgery For Painful Shoulder Osteoarthritis
Brief Title: CAM Procedure With BMAC for Shoulder OA
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of enrollment and funding for study.
Sponsor: Shane A. Shapiro (Other)
Responsible Party: Sponsor-Investigator, Shane A. Shapiro, Regulatory Sponsor, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-007731
Record Dates: First submitted 2021-03-23; First posted 2021-04-01 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Shoulder Osteoarthritis
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Subjects with Osteoarthritis of the shoulders (Experimental): Subjects diagnosed with Osteoarthritis of the shoulders will be injected with concentrated bone marrow aspirate administration after Comprehensive Arthroscopic Management (CAM) surgical procedure.
  Interventions: Biological: Concentrated bone marrow aspirate administration after Comprehensive Arthroscopic Management (CAM) surgical procedure.

INTERVENTIONS:
Biological: Concentrated bone marrow aspirate administration after Comprehensive Arthroscopic Management (CAM) surgical procedure. — Bone marrow aspirate concentrate contains a median nucleated cell count of 121,700/uL, and platelets of 384,000/uL. This leads to a cellular dose of approximately 400 million cells.

SUMMARY:
Researchers want to find out more about the side effects of Bone Marrow Aspirate Concentrate (BMAC) and what doses of BMAC are safe for people.

ELIGIBILITY:
Inclusion Criteria

* Male and Female subjects.
* Subjects must be 50 years of age or older.
* Subjects must have OA in a single or bilateral shoulder(s) with an inferior osteophyte measuring <7 mm.
* > 1 mm joint space width in the study shoulder.
* ASES score of 14.1 to 88.5
* Osteoarthritis must be primary. Subjects must have previously tried 6 months of one of the following conservative treatments: activity modification, physical therapy, and anti-inflammatory or injection therapy.
* Patients can provide written informed consent after the nature of the study is fully explained.

Exclusion Criteria

* Patients with clinically significant abnormal hematology, serum chemistry, or urinalysis screening laboratory results. If the laboratory reports a single, non-clinically relevant, non-life-threatening result for any of these studies and is the only excluding factor it may be repeated 1 week later if the patient wishes. If the laboratory reports a single, non-clinically relevant, non-life-threatening result for any of these studies and is the only excluding factor it may be repeated 1 week later if the patient wishes. Normalization of that laboratory study will then be considered non-exclusionary. If repeat non-clinically relevant, non-life-threatening results do not normalize the patient may be further evaluated by a specialist or primary care provider to determine if lab result should be exclusionary.
* Patients taking anti-inflammatory medications (prescription or over-the-counter), including herbal therapies, within 14 days of baseline visit.
* Walch Type B2/C glenoid.
* Patients taking anti-rheumatic disease medication (including methotrexate or other antimetabolites) within the 3 months prior to study entry.
* Patients receiving injections to the treated shoulder within 3 months prior to study entry,
* Patients who are pregnant or currently breast-feeding children. Females of childbearing potential must have a negative pregnancy test prior to receiving the study drug and will agree use adequate contraception (hormonal or barrier method or abstinence) from the time of screening to a period of 3 months following completion of the drug treatment cycle. Females of childbearing potential are defined as premenopausal and not surgically sterilized, or post-menopausal for fewer than 2 years. A urine pregnancy test will be performed prior to the administration of the study drug to confirm negative results. If the urine pregnancy test is positive, the study drug will not be administered and the result will be confirmed by a serum pregnancy test. Serum pregnancy tests will be performed at a central clinical laboratory, whereas urine pregnancy tests will be performed by qualified personnel using kit.
* Patients with systemic, rheumatic or inflammatory disease of the shoulder or chondrocalcinosis, hemochromatosis, inflammatory arthritis, arthropathy of the shoulder associated with juxta-articular Paget's disease, ochronosis, hemophilic arthropathy, infectious arthritis, villonodular synovitis, and synovial chondromatosis.
* Patients with ongoing infectious disease, including HIV and hepatitis.
* Patients with clinically significant cardiovascular, renal, hepatic, endocrine disease, cancer, or diabetes.
* Patients participating in a study of an experimental drug or medical device within 30 days of study entry.
* Patients with hardware or implants in the affected shoulder.
* Patients with previous open shoulder surgery or an arthroscopic procedure requiring structural repair with anchors and/or sutures.
* Presence of large glenoid cysts
* Opiate use within three months.
* Patients taking Coumadin or Plavix

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2025-08-21 (Actual); Study Completion 2025-08-21 (Actual)

PRIMARY OUTCOMES:
Adverse Reactions | 1-3 Weeks Post-Procedure
  Occurrence of adverse reactions to BMAC when delivered after shoulder CAM procedure
Morbidity related to bone marrow aspirations from iliac crests | 1-3 Weeks Post-Procedure
  Occurrence of adverse reactions to bone marrow aspirations from iliac crests

SECONDARY OUTCOMES:
Change in Visual Analog Scale (VAS) | Screening, pre-operatively, pre-injection and at 1 week, 6 weeks, 3 months, 6 months and 12 months following surgery
  Measured using the VAS questionnaire: a validated, subjective measure for pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" (0) and "worst pain" (10).
Change in American Shoulder and Elbow Surgeons Shoulder Score (ASES) | Screening, pre-operatively, pre-injection and at 1 week, 6 weeks, 3 months, 6 months and 12 months following surgery.
  Measured using the self-reported ASES questionnaire that combines pain and activities of daily living (ADL) scores for a total score out of 100, where a higher score indicates a better outcome.
Change in Subjective Shoulder Value | Screening, pre-operatively, pre-injection and at 1 week, 6 weeks, 3 months, 6 months and 12 months following surgery
  Subjective Shoulder Value (SSV) is a single-item self-completed measure in which patients are asked to grade their shoulder as a percentage of an entirely normal shoulder, which would score 100%.
Change in range of motion | Screening, pre-operatively, pre-injection and at 1 week, 6 weeks, 3 months, 6 months and 12 months following surgery
  Measured in degrees
To collect and explore pre and post injection measures of cartilage status in the affected shoulder. | 12 Months
  Assessment of structural changes of the shoulder on conventional radiographs including measurement of inferior humeral osteophyte and joint space width

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Schoch, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials